CLINICAL TRIAL: NCT04154592
Title: The Effect of Humeral Head Depressor Muscle Co-Activation Training on Functional Outcomes in Patients Undergoing Arthroscopic Shoulder Surgery After Middle-Size Rotator Cuff Muscle Tear
Brief Title: The Effect of Humeral Head Depressor Muscle Co-Activation Training in Terms of Functional Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Caner Karartı, Caner Karartı, Hacettepe University, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019500
Record Dates: First submitted 2019-11-05; First posted 2019-11-06 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2019-11

CONDITIONS: Rotator Cuff Tears; Surgery
Keywords: rotator cuff; tear; rehabilitation
MeSH Terms: conditions — Rotator Cuff Injuries; Lacerations | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Care Provider
Masking Description: Single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): In addition to the conservative treatment of the control group, humeral head depressor muscle co-activation training will be applied for 14 weeks.
  Interventions: Other: Humeral Head Depressor Muscle Co-Activation Training- Experimental Group
- Control Group (Active Comparator): The American Society of Shoulder and Elbow Therapists' consensus statement on rehabilitation following arthroscopic rotator cuff repair will be used as guideline for rehabilitation of patients (Thigpen, C. A., Shaffer, M. A., Gaunt, B. W., Leggin, B. G., Williams, G. R., & Wilcox III, R. B. (2016). The American Society of Shoulder and Elbow Therapists' consensus statement on rehabilitation following arthroscopic rotator cuff repair. Journal of shoulder and elbow surgery, 25(4), 521-535.).
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Humeral Head Depressor Muscle Co-Activation Training- Experimental Group — In addition to the conservative treatment, humeral head depressor muscle co-activation training will be applied for 14 weeks. Participants in the coactivation group will perform the glenohumeral exercises while recruiting the pectoralis major, latissimus dorsi, and teres major muscles. To achieve this, voluntary recruitment of the pectoralis major, latissimus dorsi, and teres major will be taught prior to the demonstration of the glenohumeral exercises using visual feedback provided by EMG Biofeedback. When recruitment is correctly executed (50% of the maximum voluntary contraction signal), it should be maintained while performing the glenohumeral exercises. This will be confirmed by visualizing EMG signals during the exercise training session. During each appointment with the therapist, participants will be evaluated on their capacity to achieve the exercises while performing co-activation.
  Arms: Experimental Group
Other: Control Group — The American Society of Shoulder and Elbow Therapists' consensus statement on rehabilitation following arthroscopic rotator cuff repair will be used as guideline for rehabilitation of patients (Thigpen, C. A., Shaffer, M. A., Gaunt, B. W., Leggin, B. G., Williams, G. R., & Wilcox III, R. B. (2016). The American Society of Shoulder and Elbow Therapists' consensus statement on rehabilitation following arthroscopic rotator cuff repair. Journal of shoulder and elbow surgery, 25(4), 521-535.).
  Individuals in the control group will use shoulder straps for 6 weeks after arthroscopic shoulder surgery. These patients will be referred to physiotherapy clinics 6th week. Patients between 6 and 20 weeks (a total of 14 weeks) will be admitted to the rehabilitation program according to the guideline mentioned above.
  Arms: Control Group

SUMMARY:
Recent systematic reviews, and meta-analyses concluded that rotator cuff and scapular strengthening exercises should be included in rehabilitation programs for patients with middle-size rotator cuff muscle tear. Superior translation of the humeral head is one of the factors adversely affecting this rehabilitation process. Aside from rotator cuff muscles, opposition of superior humeral head translation can be achieved by the glenohumeral adductors (i.e. pectoralis major, latissimus dorsi muscles, and teres major), which act as humeral head depressors by means of the medio-inferior vector created by the orientation of their tendons. Recruitment of the glenohumeral adductors has been shown to decrease subacromial narrowing in elevated arms in asymptomatic individuals, and is thought to be a coping mechanism to decrease pain in individuals with rotator cuff tear. However, to the best of our knowledge, the efficacy of humeral head depressor muscle co-activation training on functional outcomes in patients undergoing arthroscopic shoulder surgery after middle-size rotator cuff muscle tear has never been evaluated in patients with middle-size rotator cuff muscle tear. Since recruitment of those muscles could prevent a decrease in subacromial space during arm elevation, it could potentially lead to improved exercise performance, earlier benefits and better treatment outcomes compared to routine rotator cuff strengthening exercises. Thus, the aim of this study was to investigate the efficacy of the humeral head depressor muscle co-activation training on functional outcomes in patients undergoing arthroscopic shoulder surgery after middle-size rotator cuff muscle tear.

DETAILED DESCRIPTION:
Shoulder pain is one of the most common types of musculoskeletal pain syndroms in the general population as its prevalence has been estimated between 7% and 26% and its annual incidence between 0.9% and 2.5%. Rotator cuff tear is one of the most common causes of painful shoulders. Lack of coordination or weakness of scapulothoracic and scapulohumeral muscles is one of the main factors thought to lead to muscle tears in shoulder. More specifically, the inability of the scapular muscles to achieve superior rotation and posterior tilt, as well as the failure of rotator cuff muscles to counter the superior humeral head translation imposed by deltoid contraction can lead to impingement of the subacromial soft tissues while performing overhead dynamic tasks. This increases the rotator cuff tears' prevalance. Aside from rotator cuff muscles, opposition of superior humeral head translation can be achieved by the glenohumeral adductors (i.e. pectoralis major, latissimus dorsi muscles, and teres major), which act as humeral head depressors by means of the medio-inferior vector created by the orientation of their tendons. Recruitment of the glenohumeral adductors has been shown to decrease subacromial narrowing in elevated arms in asymptomatic individuals, and is thought to be a coping mechanism to decrease pain in individuals with rotator cuff tear. However, to the best of our knowledge, the efficacy of humeral head depressor muscle co-activation training on functional outcomes in patients undergoing arthroscopic shoulder surgery after middle-size rotator cuff muscle tear has never been evaluated in patients with middle-size rotator cuff muscle tear. Since recruitment of those muscles could prevent a decrease in subacromial space during arm elevation, it could potentially lead to improved exercise performance, earlier benefits and better treatment outcomes compared to routine rotator cuff strengthening exercises. Thus, the aim of this study was to investigate the efficacy of the humeral head depressor muscle co-activation training on functional outcomes in patients undergoing arthroscopic shoulder surgery after middle-size rotator cuff muscle tear.

ELIGIBILITY:
Inclusion Criteria:

* the presence of middle-sized (1-3 cm) rotator cuff muscle rupture,
* undergoing arthroscopic repair surgery,
* volunteering to participate in the study.

Exclusion Criteria:

* presence of diabetic mellitus,
* stage 3 and above according to Goutallier classification,
* presence of any contraindication for mobilization (hypermobility, trauma, inflammation, etc.),
* visual, verbal, cognitive defects (aphasia, unilateral neglect, etc.),
* the presence of any neurological problem,
* the presence of cervical disc hernia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (Pain) | 14 weeks
  The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be'. The patient is asked to mark his pain level on the line between the two endpoints. The distance between 'no pain at all' and the mark then defines the subject's pain. The 11-point numeric scale ranges from '0' representing no pain to '10' representing pain as bad as you can imagine or worst pain imaginable. We use VAS to measure patient's perceived pain intensity during activity, at rest and at sleep during the last week preceding the assessment. MCIC for pain VAS is reported to be 2 points or 30%.

SECONDARY OUTCOMES:
The Constant-Murley Score | 14 weeks
  The Constant-Murley Score is the most widely used shoulder evaluating instrument in Europe despite its limitations. The 100-point scoring scale takes into account both subjective and objective measurements and is divided into four domains (pain: 15 points; activities of daily living: 20 points; range of motion: 40 points; strength: 25 points). Minimal clinically important difference (MCID) for Constant-Murley Score is reported to be between 10.4 and 17 points.
Western Ontario Rotator Cuff Index (WORC) | 14 weeks
  WORC is a disease specific self-reported instrument for rotator cuff disease. It consists 21 visual analogue scale (VAS) items in five domains: physical symptoms (six items), sports/recreation (four items), work (four items), lifestyle (four items) and emotions (three items). All items respect quality of life (QoL) aspects that can particularly be influenced by rotator cuff injury. Each item has a possible score from 0 to 100 (100 mm VAS), and these scores are added to give a total score from 0 to 2100. A score of 0 implies no reduction in QoL, and a score of 2100 is the worst score possible. The data can be converted to a percent score by inverting the raw score and then converting it to a score out of 100 (2100 'patient WORC raw score'/21). The domains are based on the WHO definition of health. WORC is determined to have the highest ratings among all shoulder instruments. The minimally clinically important change (MCIC) for WORC is reported to be 275 points or 12.8%.
DASH Score | 14 weeks
  The DASH questionnaire is a 30-item questionnaire that assesses upper extremity-related symptoms and measures functional status at the level of disability. The questionnaire consists of three sections: Symptoms; Sport and Music; and Work. The first section is composed of 30 items. The second and third sections are an optional module for Sport and Music, and four items for Work. Each item is scored with a 5-point scale: 1, no difficulty/symptoms; 2, mild difficulty/symptoms; 3, moderate difficulty/symptoms; 4, severe difficulty/symptoms; 5, extreme difficulty/symptoms (unable to do). The result of each module is summed and transformed to obtain the DASH score ranging, for each section, from 0 (best function) to 100 (severe disability).
Oxford Shoulder Score | 14 weeks
  Oxford Shoulder Score (OSS), a 12-item scale rated on a five-point Likert scale from 0-4 (0=poor function, 4=good function). Daily pain and number of repetitions per exercise during home exercises were rated in the participants' diary.
Range of Motion | 14 weeks
  A universal goniometer will be used for measuring of range of motion (flexion, extension, elevation, abduction, external rotation, and internal rotation).

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi Evran University, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ryosa A, Kukkonen J, Bjornsson Hallgren HC, Moosmayer S, Holmgren T, Ranebo M, Boe B, Aarimaa V; ACCURATE study group. Acute Cuff Tear Repair Trial (ACCURATE): protocol for a multicentre, randomised, placebo-controlled trial on the efficacy of arthroscopic rotator cuff repair. BMJ Open. 2019 May 19;9(5):e025022. doi: 10.1136/bmjopen-2018-025022. PMID 31110087
- [Background] Boudreau N, Gaudreault N, Roy JS, Bedard S, Balg F. The Addition of Glenohumeral Adductor Coactivation to a Rotator Cuff Exercise Program for Rotator Cuff Tendinopathy: A Single-Blind Randomized Controlled Trial. J Orthop Sports Phys Ther. 2019 Mar;49(3):126-135. doi: 10.2519/jospt.2019.8240. Epub 2018 Nov 30. PMID 30501388
- [Background] Overbeek CL, Kolk A, Nagels J, de Witte PB, van der Zwaal P, Visser CPJ, Fiocco M, Nelissen RGHH, de Groot JH. Increased co-contraction of arm adductors is associated with a favorable course in subacromial pain syndrome. J Shoulder Elbow Surg. 2018 Nov;27(11):1925-1931. doi: 10.1016/j.jse.2018.06.015. Epub 2018 Sep 19. PMID 30243903